CLINICAL TRIAL: NCT01338896
Title: A Multicenter, Randomized, Double-blind, Two-way Cross-over Study to Compare the Adhesiveness of Two Different Rotigotine Patch Formulations in Subjects With Parkinson's Disease
Brief Title: Study to Compare Adhesiveness of Two Different Rotigotine Patch Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP1066; 2010-024250-11 (EudraCT Number)
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-07

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine; Neupro
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A-B (Experimental): 4 day treatment (Treatment A: Rotigotine transdermal patch 8 mg/24 h, test product PR 2.2.1 followed by Treatment B: Rotigotine transdermal patch 8 mg/24 h reference patch PR 2.1.1)
  Interventions: Drug: Rotigotine transdermal patch
- Sequence B-A (Experimental): 4 day treatment (Treatment B: Rotigotine transdermal patch 8 mg/24 h reference patch PR 2.1.1 followed by Treatment A: Rotigotine transdermal patch 8 mg/24 h, test product PR 2.2.1)
  Interventions: Drug: Rotigotine transdermal patch

INTERVENTIONS:
Drug: Rotigotine transdermal patch — 8 mg/24 h, transdermal patch 8 mg/24 h, 2 days
  Other Names: Neupro

SUMMARY:
The primary objective of the study is to compare the adhesiveness of two different patch formulations of rotigotine using patch size 40 cm2, under the assumption that both patch formulations show similar adhesiveness properties.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of idiopathic Parkinson´s disease, and continuous treatment with commercially available rotigotine transdermal patch for at least 3 months, and a stable rotigotine dose including an 8 mg/24 h patch for at least 2 weeks prior to enrollment

Exclusion Criteria:

* Subjects has previously participated in this study, failed to be screened, or has participated in another study with an investigational medicinal product (IMP) or medical device within the last 30 days or is currently participating in such
* Subject with a history of significant skin hypersensitivity to adhesives, other transdermal products or recently unsolved contact dermatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The average adhesiveness score of 2 days of 24 hours patch application as rated by the investigator (or designee) | 2 days of 24 hours patch application
  The international patch adhesiveness score

SECONDARY OUTCOMES:
Patch adhesiveness of first treatment day as rated by the investigator (or designee) 24 hours after patch application | after 24 hours of patch application
  The international patch adhesiveness score
Patch adhesiveness of second treatment day as rated by the investigator (or designee) 24 hours after patch application | after 24 hour of patch application
  The international patch adhesiveness score

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (16):
- Austria (2):
  - Innsbruck
  - Vienna
- Germany (9):
  - Alzenau in Unterfranken
  - Berlin
  - Bochum
  - Böblingen
  - Cologne
  - Gera
  - Karlstadt am Main
  - Stuttgart
  - Wolfach
- United Kingdom (5):
  - Blackpool
  - Derby
  - Liverpool
  - Newcastle upon Tyne
  - Norwich

REFERENCES:
- [Derived] Elshoff JP, Timmermann L, Schmid M, Arth C, Komenda M, Brunnert M, Bauer L. Comparison of the bioavailability and adhesiveness of different rotigotine transdermal patch formulations. Curr Med Res Opin. 2013 Dec;29(12):1657-62. doi: 10.1185/03007995.2013.841666. Epub 2013 Sep 23. PMID 24006953